CLINICAL TRIAL: NCT01739595
Title: A Randomized, Double Blind, Placebo Controlled Multi-Center Phase III Study to Evaluate Normalization of Morning Testosterone Levels in Overweight Men With Acquired Hypogonadotropic Hypogonadism and Normal Sperm Concentration
Brief Title: Phase III Study to Evaluate Morning Testosterone Normalization in Overweight Men With Secondary Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZA-302
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Androxal 12.5 mg (Experimental): Androxal (enclomiphene citrate), 12.5 mg oral capsules taken once daily
  Interventions: Drug: enclomiphene citrate
- Androxal 25 mg (Experimental): Androxal (enclomiphene citrate), 25 mg oral capsules taken once daily
  Interventions: Drug: enclomiphene citrate
- Placebo (Placebo Comparator): Placebo oral capsules taken one time daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: enclomiphene citrate — oral, capsules, taken one time daily, for 3 months
  Other Names: Androxal
  Arms: Androxal 12.5 mg; Androxal 25 mg
Drug: Placebo — Oral capsule taken one time daily for 3 months
  Other Names: Dummy
  Arms: Placebo

SUMMARY:
The purpose of ZA-302 is to determine the effects of Androxal on morning testosterone and reproductive status in younger overweight men with acquired hypogonadotropic hypogonadism (confirmed morning T<300 ng/dL) and normal sperm concentration, compared to changes with placebo. Subjects must not have previously been treated with testosterone products within the last 6 months.

DETAILED DESCRIPTION:
Protocol ZA-302 is a randomized, double-blind, placebo-controlled multi-center Phase 3 study to evaluate normalization of morning testosterone levels in overweight men with acquired hypogonadotropic hypogonadism and normal baseline sperm concentrations. The study requires 10 to 12 clinic visits (2 for eye exams), and is approximately 4 to 5½ months in duration. Subjects will be treated for 12-18 weeks. At Visit 3 (Week 6) subjects who do not achieve morning T values ≥300 ng/dL will be up-titrated to 25 mg. Placebo subjects may be sham titrated. Up-titrated subjects will receive an additional 6 weeks of treatment (18 weeks total). A schedule of procedures and assessments is displayed in Section 4. The study will enroll up to 152 male subjects, up to 114 randomized to treatment with Androxal and up to 38 randomized to placebo, in a 3:1 ratio. Subjects must not have used any prior testosterone treatments within the last 6 months.

Eligible subjects must have 2 consecutive assessments of morning T below 300 ng/dL and LH below 9.4 mIU/mL. They will provide 2 sperm samples at baseline, at least 2 days apart, another 2 after 12 weeks of treatment, and up-titrated subjects will provide an additional 2 samples at the end of treatment. After 12 weeks of treatment (V5) all subjects will undergo serial T assessment for determination of the Cavg. Safety assessments will include collection of adverse events, eye examinations, physical examinations and clinical laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight (BMI 25 to 42 kg/m2 inclusive) males age 18 to 60 inclusive
2. All clinical laboratory tests within normal ranges (any clinically significant deviation of laboratory results will require approval of sponsor)
3. Previously or concurrently diagnosed as having secondary hypogonadism characterized as having 2 consecutive morning testosterone assessments < 300ng/dL, one of which must be confirmed at Baseline.
4. LH < 9.4 mIU/mL (at Visit 1 only)
5. Sperm count ≥ 15 million per milliliter (assessed twice at least 48 hours apart)
6. Ability to complete the study in compliance with the protocol
7. Ability to understand and provide written informed consent
8. Agreement to provide a total of up to 6 semen sample in a sponsor-approved clinic on up to 6 separate occasions.

Exclusion Criteria:

1. Any prior use of testosterone treatments within the last 6 months
2. Use of spironolactone, cimetidine, Clomid, 5α-reductase inhibitors, hCG, androgen, estrogen, anabolic steroid, DHEA, or herbal hormone products during the study
3. Use of Clomid in the past year
4. Uncontrolled hypertension or diabetes mellitus based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled in the study.
5. Clinically significant abnormal findings at Screening (Visit 1) or Baseline, based on the Investigator's assessment
6. A hematocrit >54% or a hemoglobin >17 g/dL (sponsor may approve enrollment of subjects with hemoglobin up to 17.5 g/dL if the subject is at a location with a high elevation)
7. Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication.
8. Known hypersensitivity to Clomid
9. Symptomatic cataracts (nuclear sclerosis cataract or cortical cataract grade > 2 based on 0-4 scale or any trace of posterior subcapsular cataract)
10. Abnormal fundoscopy exam such as central retinal vein occlusion
11. Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study
12. Irreversibly infertile or compromised fertility (cryptorchism, Kallman Syndrome, primary hypogonadism, vasectomy, or tumors of the pituitary)
13. Current or history of breast cancer
14. Current or history of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a PSA>3.6
15. Presence or history of known hyperprolactinemia with or without a tumor
16. Chronic use of medications such as glucocorticoids
17. History of drug abuse or chronic narcotic use including methadone
18. A recent history of alcoholism or illegal substance or steroid abuse (<2 years) or presence of moderate alcohol use (>21 drinks per week)
19. Subjects with known history of HIV and/or Hepatitis C
20. Subjects with end stage renal disease
21. History of liver disease (including malignancy) or a confirmed AST or ALT >3 times the upper limit of normal
22. History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia or know history of QTc interval prolongation
23. History of cerebrovascular disease
24. History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism)
25. History of erythrocytosis or polycythemia
26. Subjects with cystic fibrosis (mutation of the CFTR gene)
27. Subjects unable to provide a semen sample in a sponsor-approved clinic
28. Enrollment in a previous Androxal study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Podolski, Study Chair — Repros Therapeutics Inc.
Locations (13):
- United States (13):
  - Coastal Clinical Research, Mobile, Alabama
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Meridien Research, Bradenton, Florida
  - All Medical Research, Cooper City, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Phase One Solutions, Miami Gardens, Florida
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Rochester Clinical Research, Rochester, New York
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Texas
  - Lone Peak Family Medicine, Draper, Utah
  - Granger Medical Clinic, Riverton, Utah

REFERENCES:
- See also: Sponsor home page — http://www.reprosrx.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Androxal 12.5 mg | Androxal 25 mg | Placebo
Started | 112 | 22 | 47
Completed | 99 | 21 | 45
Not Completed | 13 | 1 | 2
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Eligibility issue | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lab assessment | 1 | 0 | 0
Not completed — Drug discrepancy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Androxal 12.5 mg | Androxal 25 mg | Placebo | Total
Number analyzed (Participants) | 112 | 22 | 47 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.6) | 45.8 (8.6) | 43.6 (10.5) | 44.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 112 | 22 | 47 | 181
Region of Enrollment [Number; unit: participants]
  United States | 112 | 22 | 47 | 181

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Testosterone in Normal Range After Treatment
Description: Proportion (percent) of subjects with average serum concentration (Cavg) for T in the normal range (300 - 1040 ng/dL) after 12 weeks of treatment. Cavg was calculated as the numerical average of 24-hour serial testosterone assessments at 0, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours after dosing.
  If the lower limit of the 95% confidence interval for the Androxal treatment group at Week 12 is at least 67%, then the coprimary endpoint based on the Cavg for testosterone would have been achieved.
  FDA specified primary endpoint did not include comparison to placebo, thus the proportion of placebo subjects with average serum concentration (Cavg) for T in the normal range (300 - 1040 ng/dL) after 12 weeks of treatment was not calculated.
Time Frame: 3 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- Androxal Subjects Pooled: Androxal (enclomiphene citrate), 12.5 mg or 25 mg oral capsules taken once daily
  enclomiphene citrate: oral, capsules, taken one time daily, for 3 months
Arm/Group | Androxal Subjects Pooled
Number analyzed (Participants) | 134
Percentage of Subjects | 81.3 [73.9 to 87.0]

2. Primary Outcome: Change in Sperm Concentration
Description: Proportion of subjects with a 50% or greater decrease in sperm concentration from baseline after 12 weeks of treatment in Androxal treated subjects to placebo.
  The difference between the proportions (placebo minus Androxal) and corresponding 95% confidence interval was determined and compared to the equivalence limit of -20%. If the lower limit of the 95% confidence interval was greater than -20%, then Androxal would be concluded to be non-inferior to placebo in causing a 50% reduction in sperm concentrations.
Time Frame: 3 months
Population: ITT
Measure: Number; unit: percentage of subjects
Arm/Group | Androxal Subjects Pooled | Placebo
Number analyzed (Participants) | 134 | 47
percentage of subjects | 14.2 | 4.3

ADVERSE EVENTS:
Arm/Group | Androxal 12.5 mg | Androxal 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/112 | 0/22 | 0/47
Other Adverse Events (participants affected / at risk) | 21/112 | 16/22 | 10/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androxal 12.5 mg (N=112) | Androxal 25 mg (N=22) | Placebo (N=47)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Androxal 12.5 mg (N=112) | Androxal 25 mg (N=22) | Placebo (N=47)
Nausea (Gastrointestinal disorders) | 4 | 1 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2
URI (Infections and infestations) | 5 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Blood testosterone decreased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Hemoglobin increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights